CLINICAL TRIAL: NCT00625729
Title: MT2007-12 Allogeneic Natural Killer Cells With Rituximab in Patients With CD20 Positive Relapsed Non-Hodgkin Lymphoma or Chronic Lymphocytic Leukemia. Strategies to Increase Sensitivity of CLL Tumor Cells to Natural Killer Cell-Immune-Mediated Cytolysis
Brief Title: Donor Natural Killer Cell Infusion, Rituximab, Aldesleukin, and Chemotherapy in Treating Patients With Relapsed Non-Hodgkin Lymphoma or Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No patients exhibited natural killer cell expansion (primary endpoint).
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007LS064; MT2007-12 (Other: Blood and Marrow Transplantation Program); UMN-0707M13561 (Other: IRB, University of Minnesota); P01CA065493 (NIH)
Record Dates: First submitted 2008-02-26; First posted 2008-02-28 (Estimated); Results first posted 2010-07-30 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — aldesleukin; Interleukin-2; IL32 protein, human; Rituximab; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated Patients (Experimental): Patients with relapsed non-Hodgkin lymphoma or chronic lymphocytic leukemia treated with donor natural killer cells infusion, rituximab, aldesleukin and chemotherapy.
  Interventions: Biological: aldesleukin; Biological: allogeneic natural killer cells; Biological: rituximab; Drug: cyclophosphamide; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: aldesleukin — Day 0-14, 10 million international units, 3 times per week for 6 doses
  Other Names: IL-2
Biological: allogeneic natural killer cells — Day 0 infusion of cells (1.5-8 x 10^7 cells/kg).
  Other Names: Natural Killer Cells
Biological: rituximab — Administered Day -8, day -1, day +6 and day +13, intravenously (IV) 357 mg/m^2
  Other Names: Rituxan
Drug: cyclophosphamide — 60 mg/kg intravenous (IV) on Day -5.
  Other Names: Cytoxan
Drug: fludarabine phosphate — Day -6 through day -2, 25 mg/m^2 intravenous (IV)
  Other Names: Fludara

SUMMARY:
RATIONALE: Aldesleukin may stimulate natural killer cells to kill cancer cells. Treating natural killer cells with aldesleukin in the laboratory may help the natural killer cells kill more cancer cells when they are put back in the body. Giving monoclonal antibodies, such as rituximab, and chemotherapy drugs, such as fludarabine and cyclophosphamide, before a donor natural killer cell infusion helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells.

PURPOSE: This phase I/II trial is studying how well giving rituximab and chemotherapy followed by a donor natural killer cell infusion that has been treated in the laboratory with aldesleukin followed by aldesleukin works in treating patients with non-Hodgkin lymphoma or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if allogeneic natural killer (NK) cells infused following chemoimmunotherapy can be safely expanded in vivo with aldesleukin.

Secondary

* To determine if interleukin-15 production at day 0 correlates with NK cells expansion.
* To determine overall response rate at 3 months.
* To determine time to progression and overall survival.
* To characterize the quantitative and qualitative toxicities of this treatment plan.
* To determine the incidence of donor products that do not meet release criteria and the NK cell numbers infused.
* To correlate clinical response with donor/recipient KIR ligand matching status, FcG receptor 3A genotype, and NK cells phenotype and function
* To determine pharmacodynamic and pharmacogenomic markers and correlate them with NK cell expansion and disease response.

OUTLINE:

* Conditioning regimen: Patients receive rituximab intravenously (IV) over 6-8 hours on days -8, -1, 6, and 13; fludarabine IV on days -6 to -2; and cyclophosphamide IV on day -5.
* Allogeneic natural killer (NK) cell administration: Patients receive aldesleukin-activated haploidentical NK cells IV over less than 1 hour on day 0. Within 4 hours after allogeneic NK cell infusion, patients receive aldesleukin subcutaneously (SC) 3 times a week for 6 doses. Patients also receive filgrastim (G-CSF) SC beginning on day 14 and continuing until absolute neutrophil count (ANC) is > 2,500/mm³ for 2 consecutive days.

Patients who achieve a complete or partial response at 28 days are eligible for allogeneic stem cell transplantation. Patients who achieve initial response at 3 months, clinically benefit from treatment, but subsequently relapse are eligible for retreatment provided all eligibility criteria are met.

Blood samples are collected periodically for correlative laboratory studies. Patients with chronic lymphocytic leukemia (CLL) also undergo bone marrow aspiration periodically for correlative laboratory studies.

After completion of study treatment, patients are followed periodically for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years or older with a diagnosis of non-Hodgkin Lymphoma or chronic lymphocytic leukemia (NHL or CLL) and one of the following:

  * Progression of NHL following at least 2 prior chemotherapy regimens, (must contain rituximab for all NHL and fludarabine for follicular NHL) defined as:

    * failure to achieve partial remission (PR) with the last chemotherapy
    * disease progression within 6 months following last chemotherapy
  * Progression of CLL/SLL (small lymphocytic lymphoma) following at least 2 prior chemotherapy regimens (containing purine analogs ) in stage Rai III or IV or symptomatic disease.
  * Relapsed NHL or CLL following stem cell transplantation for whom the option of donor lymphocyte infusion is not available or clinically indicated (e.g. recipients of autologous or umbilical cord blood [UCB] transplants).
* Available related HLA-haploidentical (human leukocyte antigen) natural killer (NK) cell adult donor by at least Class I serologic typing
* Karnofsky performance status > 60%
* Measurable disease based on modified Response Evaluation Criteria In Solid Tumors (RECIST)
* Have acceptable organ function as defined within 28 days of enrollment:

  * Hematologic: platelets ≥ 80,000 x 10^9/L; hemoglobin ≥ 9g/dL, unsupported by transfusions; absolute neutrophil count (ANC) ≥ 1000 x 10^9/L, unsupported by granulocyte-colony stimulating factor or granulocyte-macrophage colony-stimulating factor (G-CSF or GM-CS)F for 10 days or Neulasta for 21 days - the hematologic requirements are waived for patients with inadequate counts due to known bone marrow involvement by lymphoma who are otherwise eligible
  * Renal: glomerular filtration rate (GFR) > 50 ml/min
  * Hepatic: alanine aminotransferase (ALT), aspartate aminotransferase (AST) < 3 x upper limit of normal and total bilirubin <3 mg/dl
  * Pulmonary function: >50% corrected carbon monoxide diffusing capacity (DLCO) and Forced Expiratory Volume in the first second (FEV1)
  * Cardiac: no symptoms of uncontrolled cardiac disease, left ventricular ejection fraction >40%
* Off prednisone or other immunosuppressive medications for at least 3 days prior to Day 0
* Women of childbearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care.

Exclusion Criteria:

* Pregnant or lactating. The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy. Women of childbearing age must use appropriate contraceptive method.
* Active central nervous system (CNS) lymphoma/leukemia
* Active serious infection (pulmonary infiltrates or lesions are allowed only after the appropriate diagnostic testing is negative for infection or appropriate therapy was initiated for probable infection)
* Pleural effusion - large enough to be detectable on the chest x-ray
* Allergy to rituximab or IL-2
* Human immunodeficiency virus (HIV) and associated non-Hodgkins lymphoma (NHL)
* Active concurrent malignancy (except skin cancer) requiring systemic therapy in the past 2 years
* Epstein-Barr virus (EBV) post-transplant lymphoproliferative disorder
* Positive hepatitis B surface antigen (HBsAg). If Hepatitis B core antibody (HBcAb) is positive, Hepatitis B deoxyribonucleic acid (DNA) by polymerase chain reaction (PCR) will be evaluated. Positive anti HBcAb and undetectable viral load does not exclude the patient.
* Any experimental therapy in the past 30 days

Donor Selection:

* Related donors (sibling, parent, offspring, parent or offspring of an HLA identical sibling) ≥ age 18 years
* Able and willing to undergo lymphapheresis
* HLA-haploidentical donor/recipient match. If time permits and multiple donors are available, preference will be given to the Killer-cell Immunoglobulin-like Receptors (KIR) ligand mismatched donor (as predicted by HLA typing).
* HIV-1, HIV-2 negative, Human T-lymphotropic virus Type I (HTLV-1), HTLV-2 negative, West Nile virus (WNV) negative, Hepatitis B and C negative
* Adequate organ function defined as:

  * Hematologic: CBC/diff/platelet count near normal limits,
  * Hepatic: ALT < 2 x upper limit of normal,
* Not pregnant or lactating
* In general good health as determined by the study physician
* Able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Bachanova, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Treated With Natural Killer Cells: Patients with relapsed non-Hodgkin lymphoma or chronic lymphocytic leukemia treated with 1 dose donor natural killer cells infusion, 4 doses rituximab, 6 doses aldesleukin and 5 doses fludarabine and 1 dose cyclosphosphamide.
Period: Overall Study
Arm/Group | Patients Treated With Natural Killer Cells
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Treated With Natural Killer Cells
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Exhibiting Natural Killer Cell Expansion
Description: Successful natural killer (NK) cell expansion will be defined as an absolute circulating donor-derived NK cell count of >100 cells/μl 14 days after infusion with <5% donor T and B cells in the mononuclear population.
Time Frame: Day 14
Measure: Number; unit: Participants
Arm/Group | Patients Treated With Natural Killer Cells
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Number of Patients With Interleukin-15 Production and NK Cell Expansion
Description: Correlation of interleukin-15 production at day 0 with natural killer (NK) cells expansion
Time Frame: Day 0
Population: Correlation of interleukin-15 with Natural Killer Cell expansion cannot be calculated because there was no Natural Killer Cell expansion.
Measure: Number; unit: Participants
Arm/Group | Patients Treated With Natural Killer Cells
Number analyzed (Participants) | 6
Participants | 0

3. Secondary Outcome: Number of Patients With Overall Response
Description: Overall response (complete remission plus partial remission) rate at 3 months, as defined by International Working Group for non-Hodgkin lymphoma and NCI Working Group guidelines for chronic lymphocytic leukemia
Time Frame: 3 Months
Measure: Number; unit: Participants
Arm/Group | Patients Treated With Natural Killer Cells
Number analyzed (Participants) | 6
Participants | 4

4. Secondary Outcome: Number of Patients Whose Disease Progressed After Treatment
Description: Includes patients (with non-Hodgkin leukemia or chronic lymphocytic leukemia) whose disease progressed after treatment.
Time Frame: 6 Months
Population: Only patients who responded to treatment included in the analysis.
Measure: Number; unit: Participants
Groups:
- Responder Patients: Patients with relapsed non-Hodgkin lymphoma or chronic lymphocytic leukemia treated with donor natural killer cells infusion, rituximab, aldesleukin and chemotherapy who had a response to treatment (clinical response or partial response).
Arm/Group | Responder Patients
Number analyzed (Participants) | 4
Participants | 2

5. Secondary Outcome: Number of Patients With Adequate Natural Killer Cells Infused
Description: Incidence of donor products that met release criteria in accordance with FDA regulations (Lot Release Criteria for allogeneic, interleukin-2 (IL-2) activated natural killer (NK) cell products (BB-IND 8847) and the NK cell numbers infused (donor NK cell dose 1.5-8.0 x 10^7/kg).
Time Frame: Day 0
Measure: Number; unit: Participants
Arm/Group | Patients Treated With Natural Killer Cells
Number analyzed (Participants) | 6
Participants | 6

6. Secondary Outcome: Number of Patients With Overall Survival
Description: Number of patients alive at 6 months after treatment.
Time Frame: 6 Months
Measure: Number; unit: Participants
Arm/Group | Patients Treated With Natural Killer Cells
Number analyzed (Participants) | 6
Participants | 3

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected after start of chemotherapy treatment (Day -1) through date of death (all within 6 months).
Description: Stopping Rules for excess toxicity:
  * Any non-hematologic grade 4 toxicity except for fevers alone
  * Grade III/IV GvHD or GvHD requiring more than 7 days of therapy
  * Hematologic toxicity: prolonged neutropenia defined as an absolute neutrophil count of less than 500 on day +35. Prolonged anemia or thrombocytopenia will not constitute toxicity.
Arm/Group | Patients Treated With Natural Killer Cells
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With Natural Killer Cells (N=6)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) — Ventricular arrhythmia - Bigeminy
Death - Disease Progression NOS (General disorders) | 3 (3)
Infection (Infections and infestations) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) — ANC <500 at day +35
Pulmonary - obstruction/stenosis of airway (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early due to lack of NK expansion and failure to meet primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No